CLINICAL TRIAL: NCT03861052
Title: A Phase 3 Study of Tirzepatide Monotherapy Compared to Dulaglutide 0.75 mg in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of Tirzepatide (LY3298176) Compared to Dulaglutide in Participants With Type 2 Diabetes
Acronym: SURPASS J-mono
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17077; I8F-JE-GPGO (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Results first posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide; dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 5 mg Tirzepatide (Experimental): Participants received 5 milligram (mg) tirzepatide administered subcutaneously (SC) once weekly for 52 weeks.
  Interventions: Drug: Tirzepatide
- 10 mg Tirzepatide (Experimental): Participants received 10 mg tirzepatide administered SC once weekly for 52 weeks.
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): Participants received 15 mg tirzepatide administered SC once weekly for 52 weeks.
  Interventions: Drug: Tirzepatide
- 0.75 mg Dulaglutide (Active Comparator): Participants received 0.75 mg dulaglutide administered SC once weekly for 52 weeks.
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 10 mg Tirzepatide; 15 mg Tirzepatide; 5 mg Tirzepatide
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
  Arms: 0.75 mg Dulaglutide

SUMMARY:
The reason for this study is to see if the study drug tirzepatide (LY3298176) is effective and safe compared to dulaglutide in participants with type 2 diabetes in Japan.

ELIGIBILITY:
Inclusion Criteria:

Participant must:

* Have been diagnosed with type 2 diabetes mellitus based on the World Health Organization classification before the screening visit.
* Have HbA1c meeting the following criteria, as determined by the central laboratory at screening and baseline:

  * for participants who are oral antihyperglycemic medication (OAM)-naïve at screening, ≥7.0% to ≤10.0% at both screening and baseline.
  * for participants who have been taking OAM monotherapy at screening, ≥6.5% to ≤9.0% at screening, and ≥7.0% to ≤10.0% at baseline.
* Have body mass index (BMI) of ≥23 kilograms per meter squared at screening.
* Be of stable weight (±5%) during 3 months preceding screening; and agree to not initiate an intensive diet and/or exercise program during the study with the intent of reducing body weight other than the lifestyle and dietary measures for diabetes treatment.

Exclusion Criteria:

Participant must not:

* Have type 1 diabetes mellitus.
* Have had chronic or acute pancreatitis any time prior to study entry.
* Have proliferative diabetic retinopathy or diabetic maculopathy or nonproliferative diabetic retinopathy requiring immediate or urgent treatment.
* Have disorders associated with slowed emptying of the stomach, or have had any stomach surgeries for the purpose of weight loss.
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease, or blood alanine transaminase (ALT) enzyme level >3.0 times the upper limit of normal (ULN) for the reference range, as determined by the central laboratory. Participants with nonalcoholic fatty liver disease (NAFLD) are eligible for participation in this trial only if there ALT level is ≤3.0 the ULN for the reference range.
* Have had a heart attack, stroke, or hospitalization for congestive heart failure in the past 2 months.
* Have a personal or family history of medullary thyroid carcinoma or personal history of multiple endocrine neoplasia syndrome type 2.
* Have been taking weight loss drugs, including over-the-counter medications during the last 3 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (46):
- Japan (46):
  - Akaicho Clinic, Chiba, Chiba
  - Medical corporation THY Tokuyama Clinic, Chiba Mihama-ku, Chiba
  - National Hospital Organization Kure Medical Center, Kure, Hiroshima
  - Hasegawa Medical Clinic, Chitose, Hokkaido
  - Yuri Ono Clinic, Sapporo, Hokkaido
  - Watanabe Naika Clinic, Nishinomiya, Hyōgo
  - Hayashi Clinic, Nishinomiya, Hyōgo
  - Naka Memorial Clinic, Naka, Ibaraki
  - Hayashi Diabetes Internal Medicine Clinic, Chigasaki-sh, Kanagawa
  - Matoba Diabetes Clinic, Ebina, Kanagawa
  - Takai Naika Clinic, Kamakura, Kanagawa
  - Kanto Rosai Hospital, Kawasaki, Kanagawa
  - H.E.C. Science Clinic, Yokohama, Kanagawa
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - Senrichuo Ekimae Clinic, Toyonaka, Osaka
  - Asano Clinic, Kawagoe, Saitama
  - Kawaguchi General Hospital, Kawaguchi, Saitama
  - Wakakusa Clinic, Shimotsuke, Tochigi
  - Seiwa Clinic, Adachi-ku, Tokyo
  - HDC Atlas Clinic, Chiyoda City, Tokyo
  - Meiwa Hospital, Chiyodaku, Tokyo
  - Asahi Life Foundation Adult Disease Research Center, Chuo-ku, Tokyo
  - Nihonbashi Sakura Clinic, Chuo-ku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Medical Corporation Chiseikai Tokyo Center Clinic, Chuo-ku, Tokyo
  - Tokyo aSBo Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - IHL Shinagawa East One Medical Clinic, Minato-ku, Tokyo
  - Sato Medical Clinic, Ootaku, Tokyo
  - Shinjuku Research Park Clinic, Shinjuku, Tokyo
  - Medical Corporation Heishinkai ToCROM Clinic, Shinjuku-ku, Tokyo
  - Tomonaga Clinic, Shinjuku-ku, Tokyo
  - Shinei Clinic, Suginami, Tokyo
  - Ikebukuro Metropolitan Clinic, Toshima-ku, Tokyo
  - Futata Tetsuhiro Clinic, Fukuoka
  - JR Hiroshima Hospital, Hiroshima
  - Yoshimura Clinic, Kumamoto
  - Keiseikai Kajiyama Clinic, Kyoto
  - OKAYAMA Medical Center, Okayama
  - AMC Nishiumeda Clinic, Osaka
  - Kitada Clinic, Osaka
  - Nanko Clinic, Osaka
  - Abe Clinic, Ōita
  - Suruga Clinic, Shizuoka
  - Yokohama Minoru Clinic, Yokohama

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mimura H, Oura T, Chin R, Hirase T, Shimono D. Association Between Early Weight Loss and Metabolic Outcomes with Tirzepatide in Japanese Patients with Type 2 Diabetes: A SURPASS J Post Hoc Analysis. Diabetes Ther. 2025 Sep;16(9):1871-1885. doi: 10.1007/s13300-025-01775-y. Epub 2025 Jul 25. PMID 40711720
- [Derived] Hamamoto Y, Oura T, Hirase T. Insulin Sensitivity and Beta-Cell Function Following Tirzepatide in Japanese Patients with Type 2 Diabetes: A SURPASS J-mono Analysis. Diabetes Ther. 2025 Apr;16(4):717-729. doi: 10.1007/s13300-025-01704-z. Epub 2025 Feb 14. PMID 39951042
- [Derived] Onishi Y, Oura T, Takeuchi M. Metabolic Abnormalities Following Tirzepatide Monotherapy in Japanese Patients with Type 2 Diabetes: A Phase 3 SURPASS J-mono Post Hoc Analysis. Diabetes Ther. 2024 Mar;15(3):649-661. doi: 10.1007/s13300-024-01534-5. Epub 2024 Feb 4. PMID 38310163
- [Derived] Ishii H, Oura T, Takeuchi M. Treatment Satisfaction and Quality of Life with Tirzepatide Versus Dulaglutide Among Japanese Patients with Type 2 Diabetes: Exploratory Evaluation of the SURPASS J-mono Trial. Diabetes Ther. 2023 Dec;14(12):2173-2183. doi: 10.1007/s13300-023-01485-3. Epub 2023 Oct 16. PMID 37843771
- [Derived] Inagaki N, Takeuchi M, Oura T, Imaoka T, Seino Y. Efficacy and safety of tirzepatide monotherapy compared with dulaglutide in Japanese patients with type 2 diabetes (SURPASS J-mono): a double-blind, multicentre, randomised, phase 3 trial. Lancet Diabetes Endocrinol. 2022 Sep;10(9):623-633. doi: 10.1016/S2213-8587(22)00188-7. Epub 2022 Jul 30. PMID 35914543
- [Derived] Sattar N, McGuire DK, Pavo I, Weerakkody GJ, Nishiyama H, Wiese RJ, Zoungas S. Tirzepatide cardiovascular event risk assessment: a pre-specified meta-analysis. Nat Med. 2022 Mar;28(3):591-598. doi: 10.1038/s41591-022-01707-4. Epub 2022 Feb 24. PMID 35210595

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 mg Tirzepatide: Participants received 5 mg tirzepatide administered SC once weekly for 52 weeks.
Period: Overall Study
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide
Started | 159 | 158 | 160 | 159
Received at Least One Dose of Study Drug | 159 | 158 | 160 | 159
Completed | 155 | 151 | 155 | 154
Not Completed | 4 | 7 | 5 | 5
Not completed — Adverse Event | 1 | 1 | 2 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 3 | 0
Not completed — Relocation to other city | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide | Total
Number analyzed (Participants) | 159 | 158 | 160 | 159 | 636
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 120 | 123 | 124 | 111 | 478
  >=65 years | 39 | 35 | 36 | 48 | 158
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 39 | 28 | 42 | 155
  Male | 113 | 119 | 132 | 117 | 481
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 159 | 158 | 160 | 159 | 636
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 159 | 158 | 160 | 159 | 636
Hemoglobin A1c [HbA1c] [Mean (Standard Deviation); unit: percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  percentage of HbA1c | 8.18 (0.88) | 8.19 (0.86) | 8.19 (0.89) | 8.15 (0.86) | 8.18 (0.87)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model for post-baseline measures: Variable = Baseline + Baseline BMI Group (<25 or >=25 kg/m^2) + Washout of Antidiabetic Medication + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: All randomized participants who received at least 1 dose of study drug and had a baseline and at least 1 post-baseline value, excluding data after initiating rescue antihyperglycemic medication or prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide
Number analyzed (Participants) | 158 | 156 | 159 | 159
percentage of HbA1c | -2.37 (0.066) | -2.55 (0.067) | -2.82 (0.066) | -1.29 (0.065)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -1.09, 95% CI 2-sided [-1.27 to -0.90]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -1.27, 95% CI 2-sided [-1.45 to -1.08]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -1.53, 95% CI 2-sided [-1.71 to -1.35]

2. Secondary Outcome: Percentage of Participants With HbA1c of <7.0%
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide
Number analyzed (Participants) | 158 | 156 | 159 | 159
percentage of participants | 93.67 | 96.79 | 99.37 | 67.30
Statistical Analysis 1: Comparison: 5 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 9.89, 95% CI 2-sided [4.53 to 21.55]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 20.57, 95% CI 2-sided [7.73 to 54.71]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 85.31, 95% CI 2-sided [15.80 to 460.58]

3. Secondary Outcome: Change From Baseline in Fasting Serum Glucose
Description: Fasting serum glucose (FSG) is a test to determine sugar levels in serum sample after an overnight fast. LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Baseline BMI Group (<25 or >=25 kg/m^2) + Washout of Antidiabetic Medication + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligrams per decilitre (mg/dL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide
Number analyzed (Participants) | 158 | 156 | 159 | 159
milligrams per decilitre (mg/dL) | -57.9 (1.73) | -64.6 (1.76) | -67.6 (1.75) | -31.9 (1.73)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -25.9, 95% CI 2-sided [-30.7 to -21.1]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -32.7, 95% CI 2-sided [-37.5 to -27.8]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -35.7, 95% CI 2-sided [-40.6 to 30.9]

4. Secondary Outcome: Change From Baseline in Average 7-Point Self-Monitored Blood Glucose (SMBG) Values
Description: The self-monitored plasma glucose (SMBG) data were collected at the following 7 time points: Morning Premeal - Fasting, Morning 2-hour Postmeal, Midday Premeal, Midday 2-hour Postmeal, Evening Premeal, Evening 2-hour Postmeal and Bedtime. LS mean was determined by analysis of covariance (ANCOVA) model for with Baseline + Baseline HbA1c Group (<=8.5%, >8.5%) + Baseline BMI Group (<25 or >=25 kg/m^2) + Washout of Antidiabetic Medication + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- 5 mg Tirzepatide: Participants received 5 mg tirzepatide administered SC once weekly for 52 week
- 10 mg Tirzepatide: Participants received 10 mg tirzepatide administered SC once weekly for 52 week
- 15 mg Tirzepatide: Participants received 15 mg tirzepatide administered SC once weekly for 52 week
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide
Number analyzed (Participants) | 141 | 133 | 135 | 137
mg/dL | -59.5 (1.46) | -64.2 (1.50) | -68.6 (1.50) | -42.2 (1.48)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -17.3, 95% CI 2-sided [-21.4 to -13.2]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -22.0, 95% CI 2-sided [-26.1 to -17.9]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -26.4, 95% CI 2-sided [-30.5 to -22.2]

5. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight. LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Baseline HbA1c Group (<=8.5%, >8.5%) + Washout of Antidiabetic Medication + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide
Number analyzed (Participants) | 158 | 156 | 159 | 159
kilogram (kg) | -5.8 (0.41) | -8.5 (0.42) | -10.7 (0.41) | -0.5 (0.41)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -5.2, 95% CI 2-sided [-6.4 to -4.1]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -7.9, 95% CI 2-sided [-9.1 to -6.8]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -10.1, 95% CI 2-sided [-11.3 to -9.0]

6. Secondary Outcome: Percentage of Participants Who Achieve Weight Loss ≥5% From Baseline
Description: Percentage of participants who achieve weight loss ≥5% from baseline.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide
Number analyzed (Participants) | 158 | 156 | 159 | 159
percentage of participants | 60.76 | 82.05 | 89.31 | 10.69
Statistical Analysis 1: Comparison: 5 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 14.44, 95% CI 2-sided [7.88 to 26.46]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 44.96, 95% CI 2-sided [23.12 to 87.45]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 82.67, 95% CI 2-sided [39.84 to 171.52]

7. Secondary Outcome: Change From Baseline in Fasting Insulin
Description: Fasting Insulin is a test used to measure the amount of insulin in the body. LS mean was determined by MMRM model for post-baseline measures with log (Actual Measurement) = log (Baseline) + Baseline HbA1c Group (<=8.5%, >8.5%) + Baseline BMI Group (<25 or >=25 kg/m^2) + Washout of Antidiabetic Medication + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milliunits per litre (mU/L)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide
Number analyzed (Participants) | 148 | 146 | 157 | 155
milliunits per litre (mU/L) | -1.07 (0.374) | -1.87 (0.344) | -2.00 (0.335) | 1.40 (0.482)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -2.47, 95% CI 2-sided [-3.67 to -1.28], Standard Error of Mean 0.610
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -3.27, 95% CI 2-sided [-4.43 to -2.11], Standard Error of Mean 0.592
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -3.40, 95% CI 2-sided [-4.55 to -2.25], Standard Error of Mean 0.587

8. Secondary Outcome: Change From Baseline in Fasting C-Peptide
Description: Fasting C-peptide is a test used to measure the amount of C-peptide in the body. A high level of C-peptide can mean that body is making too much insulin. LS mean was determined by MMRM model for post-baseline measures: log (Actual Measurement) = log (Baseline) + Baseline HbA1c Group (<=8.5%, >8.5%) + Baseline BMI Group (<25 or >=25 kg/m^2) + Washout of Antidiabetic Medication + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: micrograms per liter (ug/L)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide
Number analyzed (Participants) | 148 | 146 | 157 | 155
micrograms per liter (ug/L) | -0.25 (0.045) | -0.39 (0.042) | -0.37 (0.042) | 0.01 (0.052)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -0.26, 95% CI 2-sided [-0.40 to -0.13], Standard Error of Mean 0.069
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -0.40, 95% CI 2-sided [-0.53 to -0.27], Standard Error of Mean 0.067
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -0.38, 95% CI 2-sided [-0.51 to -0.25], Standard Error of Mean 0.067

9. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment B (HOMA-2B, Insulin)
Description: HOMA-2B is an estimated steady state beta cell function based on updated HOMA2 model. The HOMA2 model estimates steady state pancreatic beta cell function (%B) as a percentage of a normal reference population using simultaneously measured fasting plasma glucose and fasting insulin. LS mean was determined by MMRM model for post-baseline measures: log(Actual Measurement/Baseline) = log(Baseline) + Baseline HbA1c Group (<=8.5%, >8.5%) + Baseline BMI Group (<25 or >=25 kg/m^2) + Washout of Antidiabetic Medication + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of insulin sensitivity
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide
Number analyzed (Participants) | 146 | 137 | 147 | 153
percentage of insulin sensitivity | 38.5 (2.15) | 43.0 (2.38) | 46.3 (2.44) | 22.4 (1.66)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = 16.1, 95% CI 2-sided [10.7 to 21.4], Standard Error of Mean 2.72
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = 20.6, 95% CI 2-sided [14.9 to 26.3], Standard Error of Mean 2.90
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = 23.9, 95% CI 2-sided [18.1 to 29.7], Standard Error of Mean 2.95

10. Secondary Outcome: Change From Baseline in HOMA-2S (Insluin)
Description: HOMA2-S is an estimated insulin sensitivity based on updated HOMA2 model. The HOMA2 model is a computer model that estimates insulin sensitivity (%S) as percentages of a normal reference population using simultaneously measured fasting plasma glucose and fasting insulin. LS mean was determined by MMRM model for post-baseline measures: log(Actual Measurement) = log(Baseline) + Baseline HbA1c Group (<=8.5%, >8.5%) + Baseline BMI Group (<25 or >=25 kg/m^2) + Washout of Antidiabetic Medication + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of insulin sensitivity
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide
Number analyzed (Participants) | 146 | 137 | 147 | 153
percentage of insulin sensitivity | 14.5 (3.38) | 21.6 (3.83) | 25.7 (3.95) | -5.4 (2.52)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = 19.9, 95% CI 2-sided [11.7 to 28.2], Standard Error of Mean 4.22
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = 27.0, 95% CI 2-sided [18.0 to 36.0], Standard Error of Mean 4.59
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = 31.2, 95% CI 2-sided [22.0 to 40.4], Standard Error of Mean 4.68

11. Secondary Outcome: Rate of Hypoglycemia With Glucose < 54 mg/dL or Severe Hypoglycemia
Description: The hypoglycemia events were defined by participant reported events with blood glucose <54mg/dL) (<3.0 mmol/L] or severe hypoglycemia. Severe hypoglycemia is defined as an episode with severe cognitive impairment requiring the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma. The rate of postbaseline hypoglycemia was estimated by negative binomial model for post-baseline comparisons between treatment and control group: number of episodes = baseline hypoglycemia incidence + baseline BMI Group (<25 or >=25 kg/m^2) + washout of antidiabetic medication + baseline hemoglobin A1C (%) + treatment, with log (exposure in days/365.25) as an offset variable.
Time Frame: Baseline through Week 52
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Episodes/participant/365.25 days
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide
Number analyzed (Participants) | 159 | 158 | 160 | 159
Episodes/participant/365.25 days | 0 | 0 | 0.012 | 0

12. Secondary Outcome: Number of Participants With Anti-Tirzepatide Antibodies
Description: Number of participants with anti-tirzepatide antibodies. A participant is treatment emergent (TE) anti-drug antibody (ADA) evaluable if there is at least one non-missing test result for tirzepatide ADA for each of the baseline period and the postbaseline period. All percentages are relative to the total number of TE ADA evaluable participants in each treatment group. A TE ADA evaluable participant is considered to be TE ADA+ if the participant has at least one postbaseline titer that is a 4-fold or greater increase in titer from baseline measurement.
Time Frame: Baseline through Week 52
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide
Number analyzed (Participants) | 158 | 158 | 160 | 159
participants | 97 | 102 | 123 | 8

ADVERSE EVENTS:
Time Frame: Baseline through Week 52
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 0.75 mg Dulaglutide
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/158 | 0/160 | 0/159
Serious Adverse Events (participants affected / at risk) | 8/159 | 10/158 | 7/160 | 14/159
Other Adverse Events (participants affected / at risk) | 131/159 | 121/158 | 134/160 | 120/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=159) | 10 mg Tirzepatide (N=158) | 15 mg Tirzepatide (N=160) | 0.75 mg Dulaglutide (N=159)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sars-cov-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellopontine angle tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/113 (0) | 2/119 (2) | 0/132 (0) | 1/117 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=159) | 10 mg Tirzepatide (N=158) | 15 mg Tirzepatide (N=160) | 0.75 mg Dulaglutide (N=159)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 1 (10) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Conjunctival deposit (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Corneal disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dark circles under eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Optic disc haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 10 (35) | 11 (11) | 16 (89) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 6 (6) | 4 (4) | 7 (8) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 2 (6) | 7 (10) | 3 (4)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 4 (4) | 4 (4) | 2 (2)
Anal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 24 (28) | 28 (34) | 22 (32) | 17 (21)
Defaecation disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 27 (45) | 14 (27) | 18 (37) | 11 (20)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 9 (10) | 8 (9) | 10 (13) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 7 (8) | 3 (3)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Lumbar hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 19 (77) | 31 (67) | 32 (102) | 12 (13)
Neurogenic bowel (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic duct dilatation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (16) | 8 (17) | 19 (40) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (25) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hunger (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Injection site eczema (General disorders) | 0 (0) | 1 (22) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 2 (43) | 3 (16) | 1 (15)
Injection site hypersensitivity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (8)
Injection site oedema (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 2 (3) | 2 (46) | 3 (23) | 3 (46)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (4)
Injection site reaction (General disorders) | 2 (47) | 5 (44) | 9 (129) | 12 (80)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (9)
Malaise (General disorders) | 3 (6) | 6 (12) | 3 (4) | 3 (5)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (2) | 3 (3) | 2 (3)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0) | 6 (6) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (2)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 7 (7) | 1 (1) | 0 (0) | 2 (3)
Dermatitis infected (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 9 (9) | 2 (2) | 7 (7) | 4 (5)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 4 (4) | 2 (2) | 4 (4)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 29 (41) | 25 (28) | 22 (26) | 26 (30)
Oral herpes (Infections and infestations) | 1 (1) | 2 (2) | 1 (2) | 1 (2)
Otitis externa (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 3 (3) | 7 (9) | 6 (6) | 7 (8)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Purulence (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2) | 3 (5) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Chillblains (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 5 (6) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 8 (13) | 3 (3) | 5 (6) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Blood insulin decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carcinoembryonic antigen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 1 (5) | 1 (1) | 0 (0) | 0 (0)
Hepatitis e antibody positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insulin c-peptide decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 12 (18) | 7 (7) | 10 (14) | 5 (7)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nutritional condition abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Occult blood (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic enzymes increased (Investigations) | 1 (1) | 0 (0) | 5 (5) | 3 (4)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salmonella test positive (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 2 (2) | 5 (5) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 22 (25) | 21 (31) | 35 (107) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 9 (9)
Hyperlipasaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 3 (3) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5) | 9 (10) | 7 (8)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 4 (4) | 3 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/113 (0) | 1/119 (1) | 0/132 (0) | 0/117 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (13) | 4 (4) | 7 (8) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (32) | 8 (15) | 2 (4) | 6 (8)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple system atrophy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (12) | 1 (1) | 0 (0)
Patient elopement (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Taste disorder (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Device physical property issue (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/113 (0) | 0/119 (0) | 1/132 (1) | 1/117 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/46 (0) | 0/39 (0) | 0/28 (0) | 1/42 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0/113 (0) | 1/119 (1) | 1/132 (1) | 0/117 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/46 (0) | 0/39 (0) | 1/28 (1) | 0/42 (0)
Prostatitis (Reproductive system and breast disorders) | 1/113 (1) | 0/119 (0) | 0/132 (0) | 0/117 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (16) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Asteatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 5 (5) | 4 (4)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (15) | 1 (3)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1) | 0 (0) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 2 (2) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (7) | 2 (2) | 4 (4) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Open reduction of fracture (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 5 (5)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Internal haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (4):
  • Study Protocol: Clinical Study Protocol Amendment Version (a) (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT03861052/Prot_000.pdf
  • Study Protocol: Clinical Study Protocol Addendum Version (1) (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT03861052/Prot_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Version 2 (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT03861052/SAP_002.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Addendum Version 2 (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT03861052/SAP_003.pdf